CLINICAL TRIAL: NCT02189031
Title: Sensory Feedback Tactor Systems for Implementation of Physiologically Relevant Cutaneous Touch and Proprioception With Prosthetic Limbs
Brief Title: Sensory Feedback for Touch and Proprioception With Prosthetic Limbs
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Louis Stokes VA Medical Center (U.S. Federal Agency)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); National Institutes of Health (NIH) (NIH); The Cleveland Clinic (Other); HDT Global (Unknown); University of Alberta (Other); Shirley Ryan AbilityLab (Other); Defense Advanced Research Projects Agency (U.S. Federal Agency)
Responsible Party: Principal Investigator, Paul Marasco, Director of Amputee Research, Louis Stokes VA Medical Center
Other Study IDs: 11061-H39; R01NS081710-01 (NIH)
Record Dates: First submitted 2014-07-08; First posted 2014-07-14 (Estimated); Last update posted 2023-11-21 (Actual); Status verified 2023-03

CONDITIONS: Prosthetic
Keywords: Upper limb Amputee; Targeted Muscle Reinnervation; Prosthetic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Upper Extremity Amputee: Robust custom tactor to facilitate embodiment and proprioception
  Interventions: Device: Tactor array
- Able Bodied: Bypass tactor
  Interventions: Device: Bypass Tactor

INTERVENTIONS:
Device: Tactor array
  Groups: Upper Extremity Amputee
Device: Bypass Tactor
  Groups: Able Bodied

SUMMARY:
Upper limb amputation is a devastating injury that leaves many thousands of typically young and active individuals in the US to rely on artificial arms and hands to help restore their lost function. The investigators research is focused on helping these individuals to feel where their prosthetic limbs are moving without having to look at them by developing devices and approaches to provide sensory feedback of limb movement through the nerves that once served the missing limb.

DETAILED DESCRIPTION:
In the investigators research the investigators seek to understand the organization and (function/operation) of sensory neural systems in order to develop methods for restoring function to injured populations. One of the primary focus areas of the investigators research is working to integrate physiologically relevant sensory feedback with prosthetic limbs. To this end the investigators employ a variety of approaches that interweave disciplines such as electrophysiology, psychophysics, biomedical engineering and cognition. The investigators research team is composed of an interconnected and communicative network of clinicians, engineers, and scientists. This helps us to provide pathways from basic science discoveries that can be used to address clinical needs with transition directly to patient care.

ELIGIBILITY:
Inclusion Criteria:

Amputee criteria:

* Must be over 18 years of age
* Must be upper extremity amputee who has undergone targeted sensory reinnervation.

Able Bodied participants:

* Must be over 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Amputees who have undergone targeted sensory reinnervation
Sampling Method: Non-Probability Sample
Enrollment: 49 (Estimated)
Dates: Start 2013-02; Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Embodiment of the Prosthetic limb | Ten months
  Visual loading for fine motor tasks,questionnaires, and residual limb temperature will be assessed after 10 months of in home every day use of a custom robust tactor array for sensory feedback.

SECONDARY OUTCOMES:
Investigate the perceptions of limb movement | 6 months
  Test how closely both targeted reinnervation amputees and able bodied study participants are able to interpret limb movement using the kinesthetic perceptual illusion and physiologically relevant kinesthetic feedback.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Marasco, PhD, Principal Investigator — Louis Stokes VA Medical Center, Cleveland Clinic Lerner Research Institute
Locations (4):
- United States (3):
  - Rehabilitation Institute of Chicago, Chicago, Illinois
  - Louis Stokes VA Medical Center, Cleveland, Ohio
  - Cleveland Clinic Lerner Research Institute, Cleveland, Ohio
- University of Alberta Glenrose Rehabilitation Hospital, Edmonton, Alberta, Canada

REFERENCES:
- See also: Related Info — http://www.aptcenter.research.va.gov/

DOCUMENTS (1):
  • Informed Consent Form (2017-09-22): https://cdn.clinicaltrials.gov/large-docs/31/NCT02189031/ICF_000.pdf